CLINICAL TRIAL: NCT02571153
Title: Effects of Low Doses of Ketamine on Postoperative Quality of Recovery After Total Intravenous Anesthesia
Brief Title: Low Doses of Ketamine and Postoperative Quality of Recovery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidade Catolica de Sao Paulo (Other)
Responsible Party: Principal Investigator, Eduardo Toshiyuki Moro, Assistant Professor, Pontificia Universidade Catolica de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PUCSP 057539/2015
Record Dates: First submitted 2015-10-02; First posted 2015-10-08 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting
Keywords: Intravenous anesthesia; Postoperative nausea vomiting; Postoperative pain; Patient satisfaction; Quality of health care; Ketamine
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Patient Satisfaction | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Saline group (Placebo Comparator): Normal saline 0.9% (5 mL)
  Interventions: Drug: Normal saline
- Ketamine 0.2 (Experimental): ketamine 0.2 mg/kg (5 mL)
  Interventions: Drug: Ketamine 0.2 mg/kg
- Ketamine 0.4 (Experimental): ketamine 0.4 mg/kg (5 mL)
  Interventions: Drug: Ketamine 0.4 mg/kg

INTERVENTIONS:
Drug: Ketamine 0.4 mg/kg — Intravenous ketamine 0.4 mg/kg after induction of anesthesia
  Arms: Ketamine 0.4
Drug: Normal saline — Intravenous normal saline 0.9% 5 mL
  Arms: Saline group
Drug: Ketamine 0.2 mg/kg — Intravenous ketamine 0.2 mg/kg after induction of anesthesia
  Arms: Ketamine 0.2

SUMMARY:
There are evidences that intraoperative administration of low doses of ketamine may contribute to control the postoperative pain by acting on the N-methyl-D-aspartate (NMDA) channel, reducing the effects related to the tolerance and hyperalgesia induced by opioids. This study aims to evaluate the effects of administration of this agent not only as an analgesic but also its role in the quality of recovery from anesthesia, which includes observation of emotional, psychological and physical aspects. Patients who were scheduled to undergo total intravenous anesthesia (TIVA) for laparoscopic cholecystectomy will be enrolled in this clinical study. After induction of anesthesia, patients will receive one of three solutions according to the randomly selected group: ketamine 0,2 mg/kg; ketamine 0,4 mg/kg or saline. In the recovery room and on the ward, data related to the presence of pain, analgesic consumption, the incidence of nausea and vomiting, dizziness or hallucinations will be recorded. The next day, the quality of recovery will be evaluated by application of the questionnaire QoR40 (Quality of Recovery Questionnaire-40).

DETAILED DESCRIPTION:
Introduction It is known that nociceptive stimuli, triggered by surgery and tissue inflammation can cause peripheral sensitization and primary hyperalgesia, increases spinal responsiveness to stimuli, whether harmful or not, due to the wind-up phenomenon, and other mechanisms, with induction central sensitization. Additionally, opioids commonly employed during general anesthesia may activate, both, the antinociceptive system and the pro-nociceptive system which can lead to acute tolerance and hyperalgesia. There is evidence that NMDA receptors are involved in the development of these changes and that low doses of ketamine (< 1mg/kg) may control of postoperative pain to bind to the receptor phencyclidine the NMDA channel and inhibit the activation of the channel by glutamate non-competitively. Recently, there has been a change in pain management, which includes the observation of non-traditional variables such as those related to the concepts of satisfaction and quality of life related to health. To this end, a growing number of authors went on to assess the opinion of patients as a way to determine the quality of recovery from anesthesia, meaning the observation not only of pain intensity, but also aspects related to emotional state, comfort and independence physical. The QoR-40 questionnaire (Quality of recovery-40), a validated instrument for this purpose, allows an objective approach of these factors that can influence the perception of the patient and allows you to compare different therapeutic ways. There are no recent data on the application of this instrument to assess the effects of giving, or not, of low doses of ketamine on the quality of recovery of patients undergoing total intravenous anesthesia.

Methods After arrival in the operating room, standard American Society of Anesthesiologists (ASA) monitors will be applied. Midazolam 0.06 mg/kg and 1% lidocaine (30 mg) will be administered intravenously immediately after venoclysis. After anesthesia induction, capnographic monitoring will be added and the neuromuscular blockade will be evaluated using acceleromyography (TOF Watch). Induction and maintenance of anesthesia will be performed as follows: remifentanil, induction dose 0.5 μg/kg/min, followed by a maintenance dose of 0.3 μg/kg/min. Propofol, initial bolus (2.0 mg/kg) followed by infusion at 4 to 6 mg/kg/h. Each patient will receive rocuronium (0.6 mg/kg) before tracheal intubation. Ventilation will be controlled by adjusting the flow volume and respiratory rate to keep the end-tidal carbon dioxid (CO2) level between 30 and 40 mmHg. In the case of inadequate depth of anesthesia (movements, sweating, tachycardia, blood pressure increase >10% of the pre-induction value), propofol infusion or sevoflurane rate will be increased (by 1%); if this was not sufficient, the remifentanil infusion rate will be also increased (by 0,1 μg/kg/min). Patients who exhibit reductions in systolic arterial pressure (SAP) greater than 30% or heart rate (HR) reductions to less than 50 bpm will be given ephedrine (10 mg) and atropine (0.5 mg), respectively. After induction patients will receive one of three intravenous solutions: ketamine 0.2 mg/kg - diluted in saline until the volume of 5 mililiters (mL) (k2 group); ketamine 0.4 mg/kg diluted in saline until the volume of 5 ml (k4 group) or 5mL of 0.9% normal saline (K0 group). Hydration will be maintained with 0.9% normal saline 2 ml/kg/h. All of the participants were given dexamethasone (8 mg) and ketoprofen (100 mg) at the onset of surgery and dimenhydrinate (30 mg), dipyrone (1 g) and morphine (0.1 mg/kg) 15 minutes prior the end of the procedure. Atropine (0.01 mg/kg) and neostigmine (0.05 mg/kg) were used to achieve T4/T1>0.9 on the TOF monitor. Extubation was performed after awakening. When stable vital signs and respiration was confirmed, all patients were transferred to the postanesthesia care unit (PACU). Data related to the occurrence of pain, nausea, vomiting, dizziness or hallucinations at the PACU will be recorded as will be the length of stay in the PACU. Pain will be assessed every 15 minutes using a 0-10 numeric pain rating scale, where zero meant no pain and 10 the worst imaginable pain. Morphine (1 to 2 mg) will be administered intravenously every 10 minutes to maintain the pain score below 4 (1 mg when the pain score was <7 and 2 mg when it was ≥7). Following discharge from the PACU (minimum stay 60 minutes and Aldrete & Kroulik index >9), all of the participants will be given ketoprofen (100 mg) every 12 hours and dipyrone (30 mg/kg, maximum 1 g) every six hours intravenously. Whenever patients judged that their analgesia was insufficient, tramadol (100 mg) will be administered intravenously at eight-hour minimum intervals as needed. Postoperative nausea and vomiting (PONV) will be treated with dimenhydrinate (30 mg) intravenously. Pain score, use of analgesics, and the occurrence of nausea, vomiting, and other complications during the hospital ward stay will be recorded.

QoR40 The quality of postoperative functional recovery will be assessed by the QoR40 questionnaire, which assesses five dimensions of recovery (physical comfort - 12 items; emotional state - 7 items; physical independence - 5 items; physiological support - 7 items; and pain - 7 items). Each item is rated on a five-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR40 ranges from 40 (poorest quality of recovery) to 200 (best quality of recovery). The QoR40 will be administered by a blind investigator 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I or II
* Patients scheduled to undergo laparoscopic cholecystectomy

Exclusion Criteria:

* Patients who refuse to participate in the study
* Patients who are not able to communicate due to alterations in the level of consciousness, or neurologic, or psychiatric disease
* Contraindication of any of the drugs used in the study
* Patients who are superobese (BMI>40)
* History of alcohol or drug dependence

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo T Moro, PhD, Principal Investigator — School of Medical and Health Sciences, Pontificial Catholic University of São Paulo - PUCSP
Locations (1):
- Santa Lucinda Hospital, Sorocaba, São Paulo, Brazil

REFERENCES:
- [Background] Xie H, Wang X, Liu G, Wang G. Analgesic effects and pharmacokinetics of a low dose of ketamine preoperatively administered epidurally or intravenously. Clin J Pain. 2003 Sep-Oct;19(5):317-22. doi: 10.1097/00002508-200309000-00006. PMID 12966258
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Background] Wu L, Huang X, Sun L. The efficacy of N-methyl-D-aspartate receptor antagonists on improving the postoperative pain intensity and satisfaction after remifentanil-based anesthesia in adults: a meta-analysis. J Clin Anesth. 2015 Jun;27(4):311-24. doi: 10.1016/j.jclinane.2015.03.020. Epub 2015 Mar 29. PMID 25824051
- [Background] Pfenninger EG, Durieux ME, Himmelseher S. Cognitive impairment after small-dose ketamine isomers in comparison to equianalgesic racemic ketamine in human volunteers. Anesthesiology. 2002 Feb;96(2):357-66. doi: 10.1097/00000542-200202000-00022. PMID 11818769
- [Background] Kissin I, Bright CA, Bradley EL Jr. The effect of ketamine on opioid-induced acute tolerance: can it explain reduction of opioid consumption with ketamine-opioid analgesic combinations? Anesth Analg. 2000 Dec;91(6):1483-8. doi: 10.1097/00000539-200012000-00035. PMID 11094005

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saline Group | Ketamine 0.2 | Ketamine 0.4
Started | 45 | 45 | 45
Completed | 39 | 37 | 43
Not Completed | 6 | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Group | Ketamine 0.2 | Ketamine 0.4 | Total
Number analyzed (Participants) | 39 | 37 | 43 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 37 | 43 | 119
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 41.8 (11.3) | 47.2 (13.3) | 44.1 (11.4) | 44.3 (12.1)
Gender [Count of Participants; unit: Participants]
  Female | 31 | 34 | 37 | 102
  Male | 8 | 3 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Quality of Postoperative Recovery Assessed by QoR-40 Questionnaire 24 Hours After Surgery
Description: Quality of postoperative functional recovery assessed by the questionnaire QoR40 The quality of postoperative functional recovery was assessed by the QoR-40 questionnaire, which assesses five dimensions of recovery (physical comfort - 12 items; emotional state - 7 items; physical independence - 5 items; physiological support - 7 items; and pain - 7 items). Each item was rated on a five-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR-40 ranges from 40 (poorest quality of recovery) to 200 (best quality of recovery). The QoR-40 was administered by a blind investigator 24 hours after surgery.
Time Frame: 24 hours
Population: Total of 152 patients were first assessed for eligibility in this study; however, 17 were excluded because they refused participation, or met any of the exclusion criteria. Thus, 135 participants were randomly allocated to the study groups. Later, 6 participants in group S, 8 in group K2, and 2 in group K4 were excluded due to protocol deviations.
Measure: Mean (80% Confidence Interval); unit: units on a scale
Arm/Group | Saline Group | Ketamine 0.2 | Ketamine 0.4
Number analyzed (Participants) | 39 | 37 | 43
units on a scale | 187.8 [177.4 to 198.2] | 189.6 [177.6 to 201.6] | 186.8 [175.5 to 198.1]

2. Secondary Outcome: Length of PACU Stay
Description: Length of stay at postanesthesia recovery room
Time Frame: During the stay at postanesthesia recovery room (about 90 to 120 minutes)
Population: Patients aged 18 to 65 years old, with an ASA physical status I or II, who would be scheduled to undergo laparoscopic cholecystectomy.
Measure: Mean (80% Confidence Interval); unit: minutes
Arm/Group | Saline Group | Ketamine 0.2 | Ketamine 0.4
Number analyzed (Participants) | 39 | 37 | 43
minutes | 82.9 [59.2 to 106.6] | 84.5 [68 to 101] | 86 [52.1 to 119.9]

3. Secondary Outcome: Occurrence of Postoperative, Nausea and Vomiting
Description: Percentage of participants with postoperative nausea and vomiting at the PACU and during the hospital ward stay
Time Frame: 24 hours
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Saline Group | Ketamine 0.2 | Ketamine 0.4
Number analyzed (Participants) | 39 | 37 | 43
percentage of participants | 30.8 | 29.7 | 39.5

4. Secondary Outcome: Occurrence of Pain at PACU Using a 0-10 Numeric Pain Rating Scale
Description: Occurrence of pain at the PACU. Average Pain will be calculated. The pain score will be evaluated using a 0-10 numeric pain rating scale, where zero mean no pain and 10 the worst imaginable pain.
Time Frame: 90 minutes postanesthesia at recovery room
Population: as for outcome 2
Measure: Mean (80% Confidence Interval); unit: units on a scale
Arm/Group | Saline Group | Ketamine 0.2 | Ketamine 0.4
Number analyzed (Participants) | 39 | 37 | 43
units on a scale | 3.8 [0.2 to 7.4] | 2.6 [0 to 5.8] | 2.8 [0 to 5.8]

5. Secondary Outcome: Morphine Consumption (mg) at PACU
Description: Morphine consumption (mg) at PACU (about 90 to 120 minutes)
Time Frame: During the stay at postanesthesia recovery room (about 90 to 120 minutes)
Population: as for outcome 2
Measure: Mean (80% Confidence Interval); unit: mg
Arm/Group | Saline Group | Ketamine 0.2 | Ketamine 0.4
Number analyzed (Participants) | 39 | 37 | 43
mg | 1.6 [0 to 3.7] | 0.9 [0 to 2.4] | 1.1 [0 to 2.7]

6. Secondary Outcome: The Severity of Postoperative Pain
Description: The severity of postoperative pain was rated the higher score of pain (NRS) during the hospital ward stay.
  Pain was evaluated using a 0-10 numeric pain rating scale (NRS), where zero meant no pain and 10 the worst imaginable pain.
Time Frame: 24 hours
Population: as for outcome 2
Measure: Mean (80% Confidence Interval); unit: units on a scale
Arm/Group | Saline Group | Ketamine 0.2 | Ketamine 0.4
Number analyzed (Participants) | 39 | 37 | 43
units on a scale | 3.2 [0.4 to 6] | 2.8 [0 to 5.5] | 3.6 [0.5 to 6.5]

7. Secondary Outcome: Percentage of Participants With Tramadol Consumption
Description: Percentage of Participants with Tramadol during the ward stay
Time Frame: 24 hours
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Saline Group | Ketamine 0.2 | Ketamine 0.4
Number analyzed (Participants) | 39 | 37 | 43
percentage of participants | 5.1 | 10.8 | 13.9

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Saline Group | Ketamine 0.2 | Ketamine 0.4
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/37 | 0/43
Other Adverse Events (participants affected / at risk) | 0/39 | 0/37 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No